CLINICAL TRIAL: NCT07252791
Title: Safety and Immunogenicity of the 20-valent Pneumococcal Conjugate Vaccine (PCV20) in Children and Adolescents With Autoimmune Rheumatic Diseases
Brief Title: Safety and Immunogenicity of PCV20 in Pediatric Patients With Autoimmune Rheumatic Diseases
Acronym: PCV20-PARD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Insituto Adolfo Lutz (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 75531023.0.0000.0068
Record Dates: First submitted 2025-08-20; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Rheumatologic Disease
Keywords: Pneumococcal Conjugate Vaccine; PCV20; Autoimmune Diseases; Pediatric Rheumatology; Immunogenicity; Vaccine Safety
MeSH Terms: conditions — Autoimmune Diseases | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARDs (Experimental): PCV20 (Prevenar 20) vaccine administered intramuscularly in 1 dose depending on age and prior vaccination history.
  Interventions: Biological: Pneumococcal Vaccine
- Healthy control (Active Comparator): PCV20 (Prevenar 20) vaccine administered intramuscularly in 1 dose depending on age and prior vaccination history.
  Interventions: Biological: Pneumococcal Vaccine

INTERVENTIONS:
Biological: Pneumococcal Vaccine — 0.5 mL intramuscular dose containing polysaccharide conjugates for 20 pneumococcal serotypes (PCV20, Prevenar 20) vaccine will be administered intramuscularly in 1 dose in patients with ARDs and healthy controls.
  Other Names: 20-valent pneumococcal conjugate vaccine

SUMMARY:
This clinical trial evaluates the immunogenicity (humoral and cellular) and safety of the 20-valent pneumococcal conjugate vaccine (PCV20) in children, adolescents, and young adults aged 2-25 years with autoimmune rheumatic diseases (ARDs). All participants will receive PCV20 according to prior vaccine history. Antibody titers, opsonophagocytic activity, cellular immune responses, and adverse events will be measured up to 6 months post-vaccination. Effects of immunosuppressive therapy and physical activity levels related vaccine response will also be assessed.

DETAILED DESCRIPTION:
ARD patients are at higher risk of pneumococcal infections due to disease-related and therapy-induced immunosuppression. Despite vaccination recommendations, immunogenicity data for PCV20 in ARD pediatric populations are lacking. This prospective phase IV study will enroll 85 patients aged 2-25 years diagnosed with juvenile idiopathic arthritis (JIA), juvenile systemic lupus erythematosus (jSLE), and juvenile dermatomyositis (JDM). All will receive PCV20 per CDC guidance. Blood samples will be collected at baseline (D0), 4 weeks (D28), and 6 months (D180). The functional opsonophagocytic activity (OPA) for specific serotypes will be analyzed. Safety will be monitored through adverse event diaries, clinical evaluations, and disease activity indices. Physical activity will be evaluated by validated questionnaires and via accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-25 years
* Diagnosis of JIA, jSLE, or JDM by validated classification criteria
* Clinically stable
* Informed consent/assent

Exclusion Criteria:

* Acute infection or fever at vaccination
* Severe allergic reaction to vaccine components
* Recent blood transfusion (<6 months)
* Other vaccine within 4 weeks prior at the time of inclusion
* Pregnancy or breastfeeding
* Prior PCV20

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion Rate After Vaccination | Day 0 to Day 28 and through 180 days
  Will be defined as ≥2-fold increase in IgG titers for ≥50% of serotypes.

SECONDARY OUTCOMES:
Opsonophagocytic Antibody Titers (OPA) | Day 0 to Day 28 and through 180 days
  Blood samples will be collected at three time points: before the first dose (D0), 4 weeks after the first dose (D28), and six months after the final dose (D180). Functional opsonophagocytic anticapsular antibodies will be quantified using 6 validated serotype-specific opsonophagocytic activity (OPA) assays. Results will be expressed as geometric mean titers (GMTs) for each serotype and the percentage of participants reaching titers equal to or above the lower limit of quantification (LLOQ).
Safety Assessment | Day 1 through Day 28
  Safety will be closely monitored, and all serious adverse events will be classified as related or unrelated to the vaccine. A standardized adverse event diary will be provided to all patients and healthy controls for recording local and systemic reactions during the 4 weeks after first dose. Local reactions include: injection site pain, redness, swelling, bruising, itching, and induration. Systemic reactions include: fever, fatigue, chills, malaise, drowsiness, loss of appetite, nausea, vomiting, diarrhea, abdominal pain, dizziness, tremors, headache, fatigue, myalgia, muscle weakness, arthralgia, pruritus, and skin rash.
Impact of PCV20 vaccination on Disease Activity on patients with JIA | Day 1 through Day 28
  To evaluate the impact of PCV20 vaccination on clinical disease activity in patients with JIA, measured using JADAS27, higher scores indicate greater disease activity.
  Unit of Measure: Score (0-57)
Impact of PCV20 vaccination on Disease Activity on patients with JSLE | Day 1 through Day 28
  To evaluate the impact of PCV20 vaccination on clinical and laboratory disease activity in patients with juvenile systemic lupus erythematosus (jSLE), assessed using the SLEDAI-2K. The score incorporates clinical and laboratory manifestations of lupus, with higher scores indicating greater disease activity.
  Unit of Measure: Score (range 0-105)
Impact of PCV20 vaccination on Disease Activity on patients with JDM | Day 1 through Day 28
  To evaluate the impact of PCV20 vaccination on clinical and laboratory disease activity in patients with juvenile dermatomyositis (JDM), assessed using the Childhood Myositis Assessment Scale (CMAS). The CMAS evaluates muscle function and endurance, with higher scores indicating better muscle strength and physical performance.
  Unit of Measure: Score (range 0-52)
Influence of Immunosuppressive Treatment | Day 0 to Day 180
  To assess the short- and long-term influence of immunosuppressive treatment on the response to PCV-20 vaccination in patients with ARDs compared to healthy controls.
Seroconversion Rates after PCV20 vaccination by Physical Activity Classification | Day 1 to 180 post-vaccination
  Proportion of participants who achieve seroconversion defined as at least a twofold increase in pneumococcal serotype-specific IgG antibody concentrations compared to baseline at Days 28 and 180 following PCV20 vaccination.
  Participants will be categorized as physically active or inactive based on World Health Organization criteria using validated methods.
Geometric Mean Titers of Pneumococcal Antibodies after PCV20 Vaccination by Physical Activity Classification | Day 1 to 180 post-vaccination
  Geometric mean titers of pneumococcal serotype-specific IgG antibodies will be quantified using multiplex Luminex assay at Days 28 and 180 after PCV20 vaccination.
  Participants will be classified as physically active or inactive according to the World Health Organization criteria, based on validated methods.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kobayashi M, Bennett NM, Gierke R, Almendares O, Moore MR, Whitney CG, Pilishvili T. Intervals Between PCV13 and PPSV23 Vaccines: Recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Morb Mortal Wkly Rep. 2015 Sep 4;64(34):944-7. doi: 10.15585/mmwr.mm6434a4. PMID 26334788
- [Background] Jensen L, Christensen AE, Nielsen S, Pedersen FK, Rosthoj S, Jorgensen CS, Poulsen A. Response to pneumococcal conjugate and polysaccharide vaccination in children with rheumatic disease. Scand J Immunol. 2022 Feb;95(2):e13118. doi: 10.1111/sji.13118. Epub 2021 Nov 22. PMID 34768311
- [Background] Aikawa NE, Franca IL, Ribeiro AC, Sallum AM, Bonfa E, Silva CA. Short and long-term immunogenicity and safety following the 23-valent polysaccharide pneumococcal vaccine in juvenile idiopathic arthritis patients under conventional DMARDs with or without anti-TNF therapy. Vaccine. 2015 Jan 29;33(5):604-9. doi: 10.1016/j.vaccine.2014.12.030. Epub 2014 Dec 29. PMID 25554240
- [Background] Aikawa NE, Campos LM, Goldenstein-Schainberg C, Saad CG, Ribeiro AC, Bueno C, Precioso AR, Timenetsky Mdo C, Silva CA, Bonfa E. Effective seroconversion and safety following the pandemic influenza vaccination (anti-H1N1) in patients with juvenile idiopathic arthritis. Scand J Rheumatol. 2013;42(1):34-40. doi: 10.3109/03009742.2012.709272. Epub 2012 Sep 20. PMID 22992045
- [Background] Aikawa NE, Campos LM, Silva CA, Carvalho JF, Saad CG, Trudes G, Duarte A, Miraglia JL, Timenetsky Mdo C, Viana VS, Franca IL, Bonfa E, Pereira RM. Glucocorticoid: major factor for reduced immunogenicity of 2009 influenza A (H1N1) vaccine in patients with juvenile autoimmune rheumatic disease. J Rheumatol. 2012 Jan;39(1):167-73. doi: 10.3899/jrheum.110721. Epub 2011 Nov 15. PMID 22089462